CLINICAL TRIAL: NCT02811952
Title: Measuring Urinary Nano Particles and Arsenic and Comparing Them to Cystoscopic Findings and Urinary Cytology in Patients Suspected With Urinary Bladder Malignancy
Brief Title: Measuring Urinary Nano Particles and Metallic Compounds in TCC Patients
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Ilan Beniamin Klein, urologist, Carmel Medical Center
Other Study IDs: CMC-15-0127-CTIL
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Bladder Cancer
Keywords: bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A urine sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- study group: Patients that need that need cystoscopy due to suspicion/known bladder malignancy.
  Interventions: Other: without intervention
- control group: Patients that need cystoscopy due to others reasons than malignancy.
  Interventions: Other: without intervention

INTERVENTIONS:
Other: without intervention — without intervention

SUMMARY:
In many of urothelial carcinoma patients, one does not find common risk factors such as smoking. The medical center is located in an industrial city with known air and water pollution. The investigators decided to check the presence of nano particles and traces of metals in urinary samples of patients known and suspected for urothelial carcinoma and compare the results to both cystoscopic and cytological findings. The patients will fill a validated epidemiological respiratory disease survey and the results will be compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

Study group :

1. Patients that need cystoscopy due to suspicion/known bladder malignancy.
2. Patients that can read, understand and sign an informed consent form.

Control group:

1. Patients that need cystoscopy due to others reasons than malignancy.
2. Patients that present to the Department of Urology for surgery unrelated to malignancy of the urinary system ( prostatectomy, Incontinence repair, circumcision, hydrocele/ varicocele repair, ureteroscopy etc).

Exclusion Criteria:

Study group:

1. Patients receiving bladder irrigations, pregnant women, children and those with impaired judgment
2. Patients with a technically improper urine test.

Control group

1. Patients receiving bladder irrigations, pregnant women, children and those with impaired judgment
2. Patients with a technically improper urine test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with bladder cancer & control group
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
levels of nano particles and arsenic in urine | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Lady Davis Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided